CLINICAL TRIAL: NCT01751373
Title: Novel Assessment and Treatment Approaches for Detecting and Facilitating Functional Improvements in Post-Stroke Spasticity With Botulinum Toxin-A
Brief Title: Assessment and Management of Post-Stroke Spasticity With Botulinum Toxin-A
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sunnybrook Health Sciences Centre (Other)
Collaborators: Allergan (Industry)
Responsible Party: Principal Investigator, Dr. George Mochizuki, Principal Investigator, Sunnybrook Health Sciences Centre
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: ALSRIIIT-01
Record Dates: First submitted 2012-12-13; First posted 2012-12-18 (Estimated); Last update posted 2015-05-20 (Estimated); Status verified 2015-05

CONDITIONS: Stroke; Muscle Spasticity
Keywords: Botulinum Toxin; Rehabilitation; Electromyography; Electroencephalography; Transcranial Magnetic Stimulation
MeSH Terms: conditions — Stroke; Muscle Spasticity | interventions — Botulinum Toxins, Type A; Therapeutics; Standard of Care

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Standard Therapy (Active Comparator): Coupling focal BoNT-A injections with a therapy program comprising of functional tasks.
  Interventions: Behavioral: Standard Therapy
- Optimal Muscle Activation Therapy (Experimental): Coupling focal BoNT-A injections with a motor training program that focuses on developing and maintaining activation patterns in the muscle treated with BoNT-A.
  Interventions: Behavioral: Optimal muscle activation therapy

INTERVENTIONS:
Behavioral: Optimal muscle activation therapy — The proposed study uses a longitudinal, within-subject, pre/post intervention, cross-over design. All participants will complete each of 4 study phases (each 12 weeks long). These include: a) focal BTX injections in combination with either Standard Therapy or Optimal Muscle Activity Therapy; b) a three-month period where no treatment is given; c) focal BTX injections in combination either Standard Therapy or Optimal Muscle Activation Therapy; d) another three-month period where no treatment is given. The order of treatment phases will be counter-balanced across participants.
  Other Names: Botulinum Toxin-A; Therapy
  Arms: Optimal Muscle Activation Therapy
Behavioral: Standard Therapy
  Arms: Standard Therapy

SUMMARY:
Within the first year after stroke, approximately 38% of stroke survivors experience an increased resistance to movement, also called spasticity. One type of treatment that is approved for stroke survivors in Canada that could reduce spasticity is the injection of Botulinum toxin (BTX) into the affected muscle. While BTX reduces spasticity, there is limited evidence to show that BTX administration leads to functional improvements. This may occur because the outcomes aren't sensitive enough to detect change, some people may have better responses to BTX, or because BTX hasn't been paired with the right exercises to improve function. The aims of this research are: i) to determine if there is a way of improving the markers that measure change in response to treatment; and ii) to identify the ideal type of exercise that should be paired with BTX to allow the drug to have it greatest effect.

There are two primary research questions: a) What are the measures that will indicate whether a person with post-stroke spasticity will benefit from BTX therapy? It is hypothesized that EMG latency and amplitude, for those who best respond to BTX, will differ from those who demonstrate a weaker response to BTX; b)What is the ideal training approach for improving muscle function in stroke survivors receiving BTX injections? It is hypothesized that a training protocol that focuses on optimizing specific muscle activation patterns will demonstrate better outcomes than a training program designed to improve function.

ELIGIBILITY:
Inclusion Criteria:

* >120 days post first ischemic stroke
* Unilateral spasticity (MAS ≥ 1) of the wrist or elbow
* >18 years of age
* Medical referral for focal BoNT-A injections
* Residual active control of the wrist or elbow

Exclusion Criteria:

* Underlying neuromuscular disorders (i.e. ALS, neuropathies, myasthenia gravis)
* Inability to provide informed consent or communicate in English
* Bilateral paresis/spasticity
* Contractures
* Prescribed anti-spastic medication

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2011-05; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Amplitude and timing of electromyographic signals (EMG) | Baseline, Month 1, Month 2, Month 3, Month 6, Month 7, Month 8, Month 9, Month 12
  Change in electrical activation patterns of the target muscle(s) (i.e. muscle receiving BTX injection) and the antagonist muscle.

SECONDARY OUTCOMES:
Motor Evoked Potential amplitude | Baseline, Month 1, Month 2, Month 3, Month 6, Month 7, Month 8, Month 9, Month 12
  To measure the change in cortical excitability associated with the intervention.
Goal Attainment Scale | Baseline, 6 Months
  Change in Goal Attainment Scale
Modified Ashworth Scale | Baseline, Month 1, Month 2, Month 3, Month 6, Month 7, Month 8, Month 9, Month 12
  Change in Modified Ashworth Scale
Modified Tardieu Scale | Baseline, Month 1, Month 2, Month 3, Month 6, Month 7, Month 8, Month 9, Month 12
  Change in Modified Tardieu Scale
Frequency and amplitude of electroencephalographic (EEG) activity | Baseline, Month 1, Month 2, Month 3, Month 6, Month 7, Month 8, Month 9, Month 12
  Measurement of event-related cortical activity

CONTACTS AND LOCATIONS:
Overall Officials: George Mochizuki, PhD, Principal Investigator — Sunnybrook Health Sciences Centre
Locations (1):
- Sunnybrook Health Sciences Centre, Toronto, Ontario, Canada